CLINICAL TRIAL: NCT06304220
Title: Comparación de Dos Modelos de PPOS Para supresión Hipofisaria en Ciclos de estimulación ovárica, Desogestrel vs Medroxiprogesterona
Brief Title: Comparison of Two PPOS Models for Pituitary Suppression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NextFertility (Industry)
Collaborators: SINAE SL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MedroGestrel
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Infertility, Female; Fertility Disorders
Keywords: Primed-progestin ovarian stimulation protocol; Quality of oocytes; Oocyte yield; Ovarian Sensitivty Index; Controlled ovarian hyperstimulation
MeSH Terms: conditions — Infertility, Female | interventions — Levonorgestrel

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, and controlled clinical study with two different progestogens: desogestrel 75 mg and medroxyprogesterone acetate 10 mg.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DSG: Desogestrel (Active Comparator): Desogestrel Cerazet® 75 mg/day orally from the first day of controlled ovarian hyperstimulation (COH) until the day of trigger with agonist (GnRH-a).
  Interventions: Drug: Cerazet
- Group MPA: Medroxyprogesterone (Active Comparator): Medroxyprogesterone acetate Progevera® 10 mg/day orally from the first day of controlled ovarian hyperstimulation (COH) until the day of trigger with agonist (GnRH-a).
  Interventions: Drug: Cerazet

INTERVENTIONS:
Drug: Cerazet — Comparation of the utilization of two distinct progestogens for pituitary suppression
  Other Names: Progevera

SUMMARY:
The scarcity of evidence regarding the interchangeable use of different progestogens poses challenges, particularly in international egg donation and fertility preservation programs where standardizing protocols is crucial for achieving consistent efficacy, efficiency, and safety outcomes. Consequently, there's a pressing need for clinical studies to assess the effects of various progestogens on clinical outcomes in controlled ovarian hyperstimulation cycles. This study, a pioneering effort, aims to compare the effects of two progestogens on oocyte performance, safety, and efficiency in an egg donation program involving young, healthy, normo-responding patients.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled clinical study comparing two different progestogens for pituitary suppression in normo-responding patients undergoing controlled ovarian hyperstimulation (COH) for egg donation. Patients will be recruited on the day they begin the egg donation program. Before inclusion, patients must meet all inclusion and exclusion criteria and provide written informed consent. Each patient will be assigned a patient code based on the treatment group they are included in. Treatment with the assigned progestogens will start on the first day of COH. The standard protocol for egg donation will be followed, including stimulation with FSHr (Puregon®), pituitary suppression with either Medroxyprogesterone acetate (Progevera®) or Desogestrel (Cerazet®), and trigger with GnRH agonist (Triptorelin acetate, Decapeptyl®) 36 hours before oocyte retrieval. Patients will continue taking the assigned progestogen throughout the COH period. Oocyte quality will be assessed based on maturity and morphology, with mature oocytes classified as normal or good quality and abnormal oocytes categorized into intracytoplasmic and extracytoplasmic abnormalities. Quality assessment will be performed by two blinded embryologists.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18-29,9 kg/m2
* Ultrasound count of antral follicles prior to COH ≥ 12 follicles
* Meeting the criteria for inclusion in the egg donation program
* Normal karyotype and no active sexually transmitted diseases
* No use of combined hormonal contraceptives one month before COH

Exclusion Criteria:

* Patients excluded from the egg donation program
* Untreated sexually transmitted diseases, positive serology for HBV, HIV, HCV
* Blood disorders, neurodegenerative/psychiatric diseases, carriers of X-linked genetic diseases, oncological diseases, endometriosis.
* Oligomenorrhea (<1 menstrual cycle in 3 months)
* Use of combined hormonal contraceptives before COH

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Total number of oocytes retrieved from follicular puncture | 5 months
  The total number of oocytes retrieved from the follicular puncture shall be counted.
Number of mature oocytes (MII) retrieved from follicular puncture | 5 months
  The number of mature oocytes (MII) recovered from the follicular puncture shall be counted.

SECONDARY OUTCOMES:
Oocyte quality variables | 5 months
  Oocyte morphology will be assessed following the standard grading system established in Next Fertility, according to the criteria mentioned above.
Ovarian sensitivity index (OSI | 5 months
  total dose of gonadotrophin used/total number of MII oocytes obtained) x 1000
Follicles | 5 months
  Number of basal antral follicles of each size at the time of starting COH, Total number of follicles on the day of the second control and Number of follicles at the time of administering the trigger.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Quintero, Study Chair — NextFertility
Locations (1):
- NextFertility, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] La Marca A, Capuzzo M. Use of progestins to inhibit spontaneous ovulation during ovarian stimulation: the beginning of a new era? Reprod Biomed Online. 2019 Aug;39(2):321-331. doi: 10.1016/j.rbmo.2019.03.212. Epub 2019 Mar 29. PMID 31138494
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Martinez F, Rodriguez-Purata J, Clua E, Garcia S, Coroleu B, Polyzos N. Ovarian response in oocyte donation cycles under LH suppression with GnRH antagonist or desogestrel progestin: retrospective and comparative study. Gynecol Endocrinol. 2019 Oct;35(10):884-889. doi: 10.1080/09513590.2019.1604662. Epub 2019 May 12. PMID 31081407
- [Background] Martinez F, Rodriguez-Purata J, Beatriz Rodriguez D, Clua E, Rodriguez I, Coroleu B. Desogestrel versus antagonist injections for LH suppression in oocyte donation cycles: a crossover study. Gynecol Endocrinol. 2019 Oct;35(10):878-883. doi: 10.1080/09513590.2019.1604661. Epub 2019 May 7. PMID 31062995
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Phillips A, Hahn DW, Klimek S, McGuire JL. A comparison of the potencies and activities of progestogens used in contraceptives. Contraception. 1987 Aug;36(2):181-92. doi: 10.1016/0010-7824(87)90013-8. PMID 3427965
- [Background] Mikkelsen AL, Lindenberg S. Morphology of in-vitro matured oocytes: impact on fertility potential and embryo quality. Hum Reprod. 2001 Aug;16(8):1714-8. doi: 10.1093/humrep/16.8.1714. PMID 11473970
- [Background] Rienzi L, Ubaldi FM, Iacobelli M, Minasi MG, Romano S, Ferrero S, Sapienza F, Baroni E, Litwicka K, Greco E. Significance of metaphase II human oocyte morphology on ICSI outcome. Fertil Steril. 2008 Nov;90(5):1692-700. doi: 10.1016/j.fertnstert.2007.09.024. Epub 2008 Feb 4. PMID 18249393
- [Background] Kazemi A, Ramezanzadeh F, Nasr-Esfahani MH. The relations between dietary antioxidant vitamins intake and oxidative stress in follicular fluid and ART outcomes. Iran J Reprod Med. 2015 Sep;13(9):533-40. PMID 26568757
- [Background] Gaskins AJ, Afeiche MC, Wright DL, Toth TL, Williams PL, Gillman MW, Hauser R, Chavarro JE. Dietary folate and reproductive success among women undergoing assisted reproduction. Obstet Gynecol. 2014 Oct;124(4):801-809. doi: 10.1097/AOG.0000000000000477. PMID 25198264